CLINICAL TRIAL: NCT04609683
Title: Introductory Non-Clinical and Clinical Trial for Measuring Hydration Levels of Healthy and Heart Failure Patients Before, During, and After an Electrophysiology (EP) Procedure
Brief Title: Measuring Hydration Levels of Healthy and Heart Failure Patients Before, During, and After an Electrophysiology (EP) Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-01233
Record Dates: First submitted 2020-10-22; First posted 2020-10-30 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydrostasis group (Experimental): 50 study subjects scheduled for an EP procedure will have AleriTM sensors on subject's bicep, forearm, or wrist, to start data collection.
  Measurements will be made from the subject for a period of approximately 1 hours prior to the EP procedure. . Measurements will continue as patient is moved to the operating room. Once the EP procedure is complete, the subject will be transferred from the operating room to a hospital room, where they will stay overnight. Measurements will be made for 3-5hours post-operation.Detailed analysis will investigate how does AleriTM data correlate with known measures such as saline volume/rate, urine production volume, USG, Blood osmolality and body weight;
  Interventions: Device: AleriTM sensors

INTERVENTIONS:
Device: AleriTM sensors — AleriTM sensors are worn on the bicep or forearm and communicates through BLETM to a mobile App. The data is sent through the mobile App to web-based system processing where PHI is calculated and sent back to the mobile App.
  The AleriTM sensor has a form factor similar to a conventional arm band, with a hockey puck shape of approximately 48mm in diameter and 15mm in thickness the AleriTM sensor is a non-significant risk (NSR) device as it does not meet the definition of significant risk device (21 CFR 812.3(m)) because it is: not an implant; is not purported or represented to support or sustain human life; its use is not of substantial importance in the diagnosis, cure, treatment, mitigation, or prevention of impairment of health; and it does not present a serious risk to the health, safety, or welfare of a subject.

SUMMARY:
Subjects will be consented to wear the AleriTM sensor prior to, during, and after an Electrophysiology Procedure. During this time, the system will measure the following parameters from subjects: HR, temperature, saline volume/rate, urine production volume, USG, BPO. Data will be retrospectively analyzed to determine if the system effectively operates under these conditions, and can effectively monitor hydration levels of subjects compared to currently available methods.

DETAILED DESCRIPTION:
Study subjects scheduled for an EP procedure who have signed an informed consent form (ICF) will be admitted to the study. Prior to the EP procedure (e.g. in a hospital room or operating room at NYU Medical Center), either an employee of NYU or Hydrostasis will place sensor on subject's bicep, forearm, or wrist, start the sensor and connect the sensor to mobile app to start data collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiac arrhythmias or other cardiac conditions that are scheduled for EP procedures.
* Subject is over 18 years of age at the time of consenting
* Subject and/or legally authorized representative is willing to undergo the informed consent process prior to enrollment in the study

Exclusion Criteria:

* Pregnant subjects
* Subjects who are participating in another clinical study that may affect the results of either study
* Subjects who are unwilling or unable to wear the sensor for a period of up to 14 hours
* Subjects who are considered by the principle investigator to be medically unsuitable for study participation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
changes in body water content before, during and after an Electrophysiology Procedure | 1 hour pre-surgery, during surgery and 3-5 hours post-surgery
  Study team will compare the hydration status (changes in body water content) as predicted by the Aleri sensor to changes in volume according to the routinely reported volume exchanges. This will be a correlation study, and as such the purpose would be to use Pearsons' correlation between the device measurement and the interval changes in fluids ingested or excreted by the patient. There is no benchmark, but rather we will be looking for statistically significant correlation for any r>.5.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Jankelson, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to Lior.Jankelson@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.